CLINICAL TRIAL: NCT01484483
Title: Breast Cancer Care (BRECC) Registry - Development of a Breast Cancer Registry to Determine the Magnitude of Breast Cancer and Current Clinical Care Patterns in Kenya
Brief Title: An Observational Study to Register the Incidence of Breast Cancer and Current Clinical Care Patterns in Kenya
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25502
Record Dates: First submitted 2011-09-19; First posted 2011-12-02 (Estimated); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study, conducted by the Kenya Society for Hematology and Oncology, will develop a Breast Cancer and Care Registry (BRECC) for Kenya. Data on demographic, clinical and pathological characteristics, treatment and clinical outcome will be collected from newly diagnosed breast cancer patients. Breast cancer patients will be recruited into this registry cohort and followed up for a period of not less than five years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer
* No previous interventional therapy for breast cancer
* Ability to provide written informed consent as per GCP and local regulations

Exclusion Criteria:

* Participation in other clinical study where the diagnosis and treatment protocol is stated prior to enrolment
* Inability to assess and follow up patient outcomes, for example quality of life due to psychiatric illness or WHO/ECOG performance status IV or worse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed breast cancer patients
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-08-08 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Incidence of breast cancer in Kenya | 5 years
Breast cancer treatment patterns (drugs/dosage/schedule) in clinical practice in Kenya | 5 years

SECONDARY OUTCOMES:
Progression-free survival | 5 years
Overall survival | 5 years
Patient demographics of breast cancer patients in Kenya | 5 years
Pathology: Prevalence of tumour types | 5 years
Correlation between risk factors and clinical outcome | 5 years
Therapy duration/compliance | 5 years
Safety: Incidence of adverse events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- University of Nairobi School of Medicine; Internal Medicine and Therapeutics, Nairobi, Kenya